CLINICAL TRIAL: NCT04041622
Title: Coeliac Disease in the Nord-Trøndelag Health Study (HUNT)
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Norwegian University of Science and Technology (Other)
Collaborators: University of Oslo (Other); Oslo University Hospital (Other); Helse Nord-Trøndelag HF (Other); University of Groningen (Other); Karolinska Institutet (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Screening
Other Study IDs: 2017/924
Record Dates: First submitted 2019-07-30; First posted 2019-08-01 (Actual); Last update posted 2025-05-25 (Actual); Status verified 2025-05

CONDITIONS: Celiac Disease
Keywords: Prevalence; General population; Diagnosis; Prognosis; Etiology; Genes
MeSH Terms: conditions — Celiac Disease; Disease | interventions — Endoscopy; Biopsy

STUDY DESIGN:
Intervention Model Description: All inhabitants of Nord-Trøndelag County, Norway, above 18 years of age are invited to participate
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Endoscopy and biopsy (Other): Participants of the HUNT study with a positive serological assay for celiac disease are invited to attain a diagnostic endoscopy with duodenal biopsies
  Interventions: Diagnostic Test: Endoscopy and biopsy

INTERVENTIONS:
Diagnostic Test: Endoscopy and biopsy — Participants with a positive celiac serology are assessed by endoscopy and duodenal biopsy

SUMMARY:
In this study, all citizen of Nord-Trøndelag County, Norway, above 20 years of age are invited to participate in a population-based health study, the HUNT study. Blood samples are drawn from the participants and assessed for celiac disease by a serological assay. Celiac disease is a chronic inflammatory disease of the small intestine due to dietary gluten in wheat, barley and rye. The diagnosis will be verified through endoscopic assessment and biopsies from the small intestinal mucosa. The aims of the study are 1) to establish the population-based prevalence of celiac disease; 2) to assess the consequences of the disease from patient reported outcomes, symptoms, deficiencies, and co-morbidity; 3) to study possible risk factors and environmental triggering events; 4) to identify genetic predictors and gene-environmental interactions.

ELIGIBILITY:
Inclusion Criteria:

* Participants of the forth round of the HUNT study

Exclusion Criteria:

* None

Min Age: 20 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 56000 (Actual)
Dates: Start 2019-06-17 (Actual); Primary Completion 2024-07-01 (Actual); Study Completion 2024-07-01 (Actual)

PRIMARY OUTCOMES:
Prevalence of celiac disease | 1 year
  the proportion of cases in the general population of Nord-Trøndelag County, Norway

CONTACTS AND LOCATIONS:
Overall Officials: Eivind Ness-Jensen, md phd, Principal Investigator — NTNU, Norwegian University of Science and Technology
Locations (1):
- Levanger Hospital, Nord-Trøndelag Hospital Trust, Levanger, Norway

REFERENCES:
- [Derived] Lukina P, Andersen IL, Eggen PT, Mjones PG, Ronne E, Bolstad N, Klaasen RA, Warren DJ, Iversen R, Hveem K, Bernklev T, Jelsness-Jorgensen LP, Pedersen L, Jonkers I, Lagergren P, Sollid LM, Lundin K, Ness-Jensen E. Coeliac disease in the Trondelag Health Study (HUNT), Norway, a population-based cohort of coeliac disease patients. BMJ Open. 2024 Jan 9;14(1):e077131. doi: 10.1136/bmjopen-2023-077131. PMID 38195172